CLINICAL TRIAL: NCT00460915
Title: Korea University Guro Hospital
Brief Title: Efficacy and Safety of Lacidipine and Amlodipine on Blood Pressure in Korean ISH Patients Aged 60 to 80 Years
Acronym: ELDER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COL109776
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2009-11

CONDITIONS: Hypertension
Keywords: Lacidipine; Amlodipine
MeSH Terms: conditions — Hypertension | interventions — lacidipine; Amlodipine

INTERVENTIONS:
Drug: Lacidipine & Amlodipine

SUMMARY:
Primary Objective -To investigate the clinical effectiveness of lacidipine and amlodipine on systolic blood pressure (SBP) in Korean ISH patients aged 60 to 80 years.

Secondary Objectives -To investigate the clinical effectiveness of lacidipine and amlodipine on diastolic blood pressure (DBP) in Korean ISH patients aged 60 to 80 years

To demonstrate the effectiveness of lacidipine and amlodipine on endothelial function through measurement of markers of inflammation.

DETAILED DESCRIPTION:
Patients will receive lacidipine 4mg and amlodipine 5mg for initial 4 weeks. If SBP is less than 140mmHg at Week 4, subjects continue to take lacidipine 4mg and amlodipine 5mg.

If SBP is ≥140mmHg at Week 4, the dose of lacidipine will be increased to 6mg and amlodipine will be increased to 10mg.

If BP is not controlled under 140mmHg at Week 8, diuretics will be added. For 12 weeks of treatment period, subjects will be visit to clinic at every 4 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 55 to 80 years of age at screening
2. The subject has been newly diagnosed as essential hypertension or not treated in the past 2 weeks. If the subject took medication in the past 2 weeks, a wash-out period of at least 2 weeks will be completed prior to performing screening (week -2) assessments
3. The subject has a mean seated SBP at screening visit ≥ 140mmHg (as measured by a mercury sphygmomanometer)
4. Isolated systolic hypertension (ISH) patient (SBP≥ 140mmHg, DBP ≤90mmHg)
5. If the subject is a female of child-bearing potential, she agrees to practice acceptable contraceptive measures during the study, and for 30 days after the last dose of study medication is taken
6. The subject has given written informed consent

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply :

  1. Mean seated SBP of > 180 mmHg at screening and during the study
  2. Known or suspected secondary hypertension
  3. The subject has anemia defined by hemoglobin concentration < 10.0 g/dL for male or female
  4. The subject has a hemoglobinopathy or peripheral vascular disease
  5. The subject has presence of clinically significant renal or hepatic disease (i.e., subjects with serum creatinine > 1.4 mg/dL;ALT, AST, total bilirubin, or alkaline phosphatase > 2.5 times the upper limit of the normal (ULN) reference range
  6. The subject has presence of unstable or severe angina, coronary insufficiency, or any congestive heart failure requiring pharmacologic treatment
  7. The subject has a chronic disease requiring intermittent or chronic treatment with oral, intravenous, or intra-articular corticosteroids (i.e., only use of topical, inhaled or nasal corticosteroids is permissible)
  8. The subject has a clinically significant abnormality identified at screening which in the judgement of the investigator makes the subject unsuitable for inclusion in the study (e.g. physical examination, or electrocardiogram etc.)
  9. Past medical history or concomitant disease of metabolic acidosis or diabetic ketoacidosis
  10. The subject has a diagnosis of cancer (other than squamous or basal cell) in the past 3 years and is currently receiving treatment for the active cancer
  11. Subject who is taking medication known to affect blood pressure
  12. Known drug or alcohol dependency within 6 months prior to screening as determined by the investigator
  13. Has taken part in a clinical trial using a marketed product, investigational drug or device within 1 month prior to screening.
  14. Hypersensitivity to any component of lacidipine and amlodipine

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean SBP at week 12

SECONDARY OUTCOMES:
Change from baseline in the mean DBP at week 12
Change from baseline in the CRP at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Hong-seog Seo, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Na JO, Seo HS, Choi CU, Lim HE, Kim JW, Kim EJ, Han SW, Rha SW, Park CG, Oh DJ; ELDER investigators. Results of a 14-Week, Multicenter, Prospective, Randomized, Open-Label, Noninferiority Clinical Trial Comparing the Antihypertensive Effect and Edema Incidence of Lacidipine and Amlodipine in Older Korean Patients with Mild-to-Moderate Hypertension. Curr Ther Res Clin Exp. 2013 Jun;74:54-61. doi: 10.1016/j.curtheres.2013.02.001. PMID 24384734